CLINICAL TRIAL: NCT00898131
Title: Specialized Program of Research Excellence (SPORE) in Breast Cancer: Tissue and Specimen Collection
Brief Title: Collecting Tissue Samples for Future Research From Women Undergoing Surgery for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI 01X1; P50CA089018 (NIH); P30CA060553 (NIH); NU-NCI-01X1; NCI-01X1; STU00023488 (Other: Northwestern University IRB#)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue from diagnostic biopsies, as well as initial or follow-up surgical procedures for the treatment or prevention of breast cancer. No extra tissue is taken, only what is left over following clinical use will be retained for banking purposes.
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Collecting and storing samples of tumor tissue from patients with breast cancer to study in the laboratory may help doctors learn more about cancer.

PURPOSE: This phase I study is collecting tissue samples for future research from women undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Collect breast tissue for future research from women undergoing surgery for breast cancer.

Secondary

* Create microarrays by tumor type for internal use by Specialized Program of Research Excellence.

OUTLINE: Tumor tissue is collected and analyzed to create microarrays by tumor type for future research studies.

PROJECTED ACCRUAL: A total of 1,250 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing surgery for breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing biopsy or surgical procedures for the diagnosis, treatment, or prevention of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2001-08; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Collect human breast tissues and associated clinical-pathologic data | At time of diagnosis, surgery, and throughout standard care and clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulesza, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States